CLINICAL TRIAL: NCT01044914
Title: Use of Clinical and Intermediate Phenotypes to Assess Response to Quetiapine: the Role of Putative Causative Genes
Brief Title: Genes, Intermediate Phenotypes and Response to Quetiapine RX
Status: Completed | Type: Observational
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Alessandro Bertolino, MD. PhD, University of Bari
Other Study IDs: 2009-013028-21
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Pharmacological treatment of schizophrenia is still characterized by a certain proportion of patients who are resistant to common antipsychotics. Variability in individual response ranges from patients who experience complete or near complete symptom remission to a subset of patients who remain treatment-refractory despite extensive drug trials over years. The investigators propose to take advantage of the simultaneous acquisition of clinical and of intermediate phenotypes to ascertain the possible contribution of SNPs within putative causative genes to response to treatment with quetiapine XR.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Diagnosis of schizophrenia using the Structured Clinical Interview for Diagnosis for the Diagnostic and Statistical Manual of Mental Disorders-Fourth Edition
* Male or female patients aged between 18 and 65 years
* Female patients of childbearing potential must be using a reliable method of contraception and have a negative urine human chorionic gonadotropin test at enrollment
* Able to understand and comply with the requirements of the study
* Patients with a cut off value for PANSS more than 75

Exclusion Criteria:

* Pregnancy or lactation
* Any DSM-IV Axis I disorder not defined in the inclusion criteria
* Patients who, in the opinion of the investigator, pose an imminent risk of suicide or a danger to self or others
* Known intolerance or lack of response to quetiapine fumarate, as judged by the investigator
* Use of any of the following cytochrome P450 3A4 inhibitors in the 14 days preceding enrollment including but not limited to: ketoconazole, itraconazole, fluconazole, erythromycin, clarithromycin, troleandomycin, indinavir, nelfinavir, ritonavir, fluvoxamine and saquinavir
* Use of any of the following cytochrome P450 inducers in the 14 days preceding enrollment including but not limited to: phenytoin, carbamazepine, barbiturates, rifampin, St. John's Wort, and glucocorticoids
* Administration of a depot antipsychotic injection within one dosing interval before randomization
* Patients treated with clozapine within 28 days before the enrollment
* Substance or alcohol dependence at enrollment (except dependence in full remission, and except for caffeine or nicotine dependence)
* Opiates, amphetamine, barbiturate, cocaine, cannabis, or hallucinogen abuse by DSM-IV criteria within 4 weeks prior to enrollment
* Medical conditions that would affect absorption, distribution, metabolism, or excretion of study treatment
* Unstable or inadequately treated medical illness (e.g. diabetes, angina pectoris, hypertension) as judged by the investigator
* Involvement in the planning and conduct of the study
* Previous enrollment or randomization of treatment in the present study
* Participation in another drug trial within 4 weeks prior to enrollment into this study or longer in accordance with local requirements
* A patient with Diabetes Mellitus
* An absolute neutrophil count of ¬1.5 x 109 per liter
* Pre-existing Organic Mental Disorder or Mental Retardation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out in a hospital unit of the psychiatric assistance system.We will recruit 100 patients with schizophrenia with recent exacerbation of psychotic symptomatology.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2009-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change from baseline in clinical symptoms assessed by PANSS scores measures based on BDNF genotype in schizophrenic patients after quetiapine XR treatment | after 56 days of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Psichiatrica - Azienda Ospedaliera Policlinico Bari, Bari, Bari, Italy